CLINICAL TRIAL: NCT03613311
Title: Prevalence Rates of Evident, Occult and no Demonstrated Urodynamic Stress Incontinence and Their Clinical and Urodynamic Findings in Women With ≥Stage II Cystocele
Brief Title: Evident, Occult and no Demonstrated USI and UDS Findings in Women With ≥Stage II Cystocele
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201805048RIN
Record Dates: First submitted 2018-07-18; First posted 2018-08-03 (Actual); Last update posted 2018-08-03 (Actual); Status verified 2018-07

CONDITIONS: Urodynamic Stress Incontinence in Severe Cystocele Women
Keywords: Cystocele; Urodynamic stress incontinence; Pad test; Urodynamic study
MeSH Terms: conditions — Cystocele

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Evident urodynamic stress incontinence(USI): Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent urodynamic studies in a medical center were reviewed. USI is noted during filling cystometry and is defined as the involuntary leakage of urine during increased abdominal pressure, in the absence of a detrusor contraction.
  Interventions: Diagnostic Test: Urodynamic study
- Occult USI: Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent urodynamic studies in a medical center were reviewed. USI is noted during filling cystometry and is defined as the involuntary leakage of urine during increased abdominal pressure, in the absence of a detrusor contraction after prolapse reduction by vaginal gauze.
  Interventions: Diagnostic Test: Urodynamic study
- ND USI: Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent urodynamic studies in a medical center were reviewed. No USI was noted in this group.
  Interventions: Diagnostic Test: Urodynamic study

INTERVENTIONS:
Diagnostic Test: Urodynamic study — Urodynamic study: including uroflowmetry, filling cystometry, voiding cystometry, and urethral pressure profile

SUMMARY:
Prevalence rates of urodynamic urinary incontinence (USI) subtypes and their related clinical and urodynamic findings in women with ≥ pelvic organ prolapse quantification stage II cystocele are important for clinical consultation, especially for occult USI. Misdiagnosis of occult USI before cystocele repair might lead to occurrence of de novo stress urinary incontinence after cystocele repair. Thus, the aim of this study was to elucidate the above findings and between-group associations.

DETAILED DESCRIPTION:
Between November 2011 and January 2017, medical records of all women with ≥stage II cystocele who underwent urodynamic studies in a medical center were reviewed. ANOVA test and post-hoc testing with bonferroni's correction were used for statistical analysis. USI is noted during filling cystometry and is defined as the involuntary leakage of urine during increased abdominal pressure, in the absence of a detrusor contraction. The recruited patients with cystocele were classified into three groups (i.e.,evident USI, occult USI and no demonstrated USI) according to pad weight results before and after prolapse reduction.

ELIGIBILITY:
Inclusion Criteria:

1. Age >20y/o
2. Cystocele > stage II
3. Complete urodynamic study

Exclusion Criteria:

1. Pregnancy
2. Urinary tract infection
3. Previous pelvic reconstruction surgery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with cystocele more than stage II
Sampling Method: Non-Probability Sample
Enrollment: 480 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Evident USI | Between November 2011 and January 2017
  USI note before reduction of prolapse
Occult USI | Between November 2011 and January 2017
  USI note after reduction of prolapse

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD